CLINICAL TRIAL: NCT07170462
Title: Effect of Cranberry in Reducing Dysbiosis in Patients With Crohn's Disease
Brief Title: Cranberry and Gut Health in Crohn's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ana Maldonado-Contreras (Other)
Responsible Party: Sponsor-Investigator, Ana Maldonado-Contreras, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00002053; Gift -The Cranberry Institute (Other Grant/Funding Number: The Cranberry Institute)
Record Dates: First submitted 2025-07-17; First posted 2025-09-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease (CD); Crohn Disease
Keywords: cranberry; dietary supplement; crohn disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cranberry (Experimental): Participants in the intervention arm will be provided with 7 servings of Cranberry whole powder per week. Participants in the intervention arm are expected to consume 1 serving per day of cranberry whole powder for 10 weeks.
  Interventions: Drug: Cranberry powder
- Placebo (Placebo Comparator): Participants in the placebo arm will be provided with 7 servings of placebo powder (placebo supplement matched in appearance and flavor) per week. Participants in the placebo arm are expected to consume a serving per day of placebo powder for 10 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Cranberry powder — Cranberry whole powder equivalent to 100 g of fresh cranberries, 525 mg total (poly)phenols), and approximately 3.6 g of fiber.
  Arms: Cranberry
Dietary Supplement: Placebo — placebo powder (9 g powder, no (poly)phenols, no fibers
  Arms: Placebo

SUMMARY:
This study is investigating whether a cranberry-based dietary supplement, rich in polyphenols and fiber, can enhance gut health in individuals with Crohn's disease. People with Crohn's disease often have an imbalance in their gut microbiome (the community of bacteria in the gut). Previous research suggests that cranberry compounds may help support beneficial gut bacteria.

In this study, adults with Crohn's disease will be randomly assigned to one of two groups: one group will receive a cranberry supplement to take once daily for 10 weeks, and the other group will receive a placebo (a supplement with no active ingredients).

All participants will be asked to complete online questionnaires and collect samples of their blood, urine, and stool at four time points over a total of 15 weeks. These samples will help researchers understand how the cranberry supplement affects the gut microbiome, inflammation, and overall health.

Participation is voluntary, and participants can withdraw from the study at any time. The results of this study may help identify new diet-based approaches to improve gut health in individuals with Crohn's disease.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial evaluates the effect of a cranberry dietary supplement-rich in polyphenols and fermentable fiber-on the gut microbiome, inflammation, and health-related quality of life in adults with Crohn's disease (CD). Crohn's disease is a chronic inflammatory bowel disease associated with significant dysbiosis (disruption of the gut microbial community), and patients often experience impaired quality of life despite medical treatment. There is growing interest in food-based strategies that may favorably impact the gut microbiota in individuals with CD. Polyphenols and fermentable fibers found in whole plant foods-especially in cranberries-have demonstrated prebiotic-like effects in preclinical and small-scale human studies.

The primary aim of this study is to determine whether daily consumption of a freeze-dried, 100% cranberry powder supplement for 10 weeks improves the gut microbiome composition. Secondary objectives include assessing changes in inflammation, gastrointestinal symptoms, and quality of life, as well as evaluating the persistence of any microbiome shifts during the follow-up period after supplement cessation.

Participants are randomized 1:1 to either the intervention group (cranberry) or a control group (placebo; matched in appearance and flavor) and will consume the assigned supplement daily for 10 consecutive weeks. The total study period for each participant is 15 weeks, which includes a 10-week intervention and a 4-week follow-up phase. Participants will be blinded to group assignment, and supplements will be pre-packaged and labeled to maintain allocation concealment.

Throughout the study, participants complete questionnaires and collect biological samples at four time points: baseline (week 0), midpoint (week 6), end of intervention (week 10), and follow-up (week 14). Study assessments include the short Crohn's Disease Activity Index (sCDAI), the short Inflammatory Bowel Disease Questionnaire (sIBDQ), and dietary evaluations. These tools are used to assess changes in disease activity, gastrointestinal symptoms, health-related quality of life, and habitual diet. Participants also report any adverse events or changes in medications daily throughout the study.

Biological samples collected include stool, urine, and capillary blood (via the Tasso™ device), obtained at each time point using home collection kits. Stool samples are used for 16S rRNA sequencing and metagenomic analysis to characterize microbiome composition and function. Urine and blood are analyzed for markers f cranberry intake. Sample return is facilitated by pre-labeled, insulated packaging with cold packs. Participants receive training materials, including video instructions and support from the study team as needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult CD patients between 18 and 65 years old.
* Women of childbearing potential will be required to use at least one form of "highly effective" contraception throughout the study.
* Confirmed diagnosis of Crohn's disease.
* CD activity lower than sCDAI<450.
* Moderate to severely impaired Health Related Quality of life (HRQoL). sIBDQ score <60.
* Stable dose of medications at screening; thiopurines, natalizumab, methotrexate (12 weeks), anti-TNF, ustekinumab (8 weeks), vedolizumab (8 weeks), 5-ASA (2 weeks),
* steroids (1 week).
* Willingness and capacity to significantly consume the cranberry supplement daily.
* Willing and able to comply with specimen collection and other study procedures, and to complete the study.
* Able to provide written informed consent.
* Reside in Massachusetts, USA.

Exclusion Criteria:

* Ostomy
* Presence of symptomatic or significant stricture or history of obstruction in the past 6 months
* Pregnancy
* Use of Specific Carbohydrate Diet of IBD- AID within 4 weeks of screening
* Use of probiotics within 4 weeks of screening
* Use of antibiotics within 4 weeks of screening
* > 20mg prednisone or equivalent
* Recent C. difficile colitis
* Unable to provide informed consent for themselves
* Prisoners
* Children

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in relative abundance of butyrate-producing Clostridia species, assessed with shotgun metagenomic sequencing and MetaPhlAn taxonomic profiling | 15 weeks
  Stool samples will be collected at Baseline and during the intervention. DNA will be extracted and sequenced using paired-end shotgun metagenomics (2×150 bp). Taxonomic profiling will be performed with MetaPhlAn to quantify species-level relative abundance. The primary endpoint is the within-participant change in the summed relative abundance (%) of butyrate-producing Clostridia (clusters IV & XIVa). For each participant, species-level abundances will be summed to create a composite (%). The primary analysis will compare mean change from Baseline to time points during the intervention between intervention and placebo groups, with results summarized as mean change and between-group differences with 95% CIs. The unit measure is relative abundance, %.

SECONDARY OUTCOMES:
Proportion of participants with ≥70-point reduction in short Crohn's Disease Activity Index (sCDAI) score | 15 weeks
  The short Crohn's Disease Activity Index (sCDAI) questionnaire will be administered at baseline and during the intervention. Scores are calculated from patient-reported symptoms and range from 0 to 600, with higher values indicating more severe disease activity. The outcome is the proportion of participants achieving at least a 70-point reduction in sCDAI score from baseline. The principal comparison is the between-group difference (cranberry intervention vs placebo) in the percentage of participants reaching this clinical response threshold.
Mean change in short Crohn's Disease Activity Index (sCDAI) score | 15 weeks
  The short Crohn's Disease Activity Index (sCDAI) will be used to assess disease activity at baseline and during the intervention. Scores range from 0 to 600, with higher scores reflecting more active Crohn's disease. The outcome is the within-participant change from baseline in sCDAI score. The primary comparison is the between-group difference (cranberry intervention vs placebo) in mean change from Baseline, reported as mean (SD) change and between-group differences with 95% confidence intervals.
Proportion of participants achieving short Crohn's Disease Activity Index (sCDAI) <150 points | 15 weeks
  The short Crohn's Disease Activity Index (sCDAI) will be assessed at baseline and during intervention. Scores range from 0 to 600, with higher scores indicating greater Crohn's disease activity. The outcome is the proportion of participants with sCDAI <150 after the intervention, which is a commonly accepted definition of clinical remission. The principal comparison is the between-group difference (cranberry intervention vs placebo) in the percentage of participants meeting this remission threshold.
Proportion of participants with ≥50% reduction in short Inflammatory Bowel Disease Questionnaire (SIBDQ) score | 15 weeks
  The short Inflammatory Bowel Disease Questionnaire (SIBDQ) will be administered at baseline and during the intervention to evaluate health-related quality of life in participants with IBD. Scores range from 10 to 70, with higher scores indicating better quality of life. The outcome is the proportion of participants who demonstrate a ≥50% reduction in their SIBDQ score from baseline. The main comparison is the between-group difference (cranberry intervention vs placebo) in the proportion of participants achieving this reduction.
Proportion of participants achieving C-reactive protein (CRP) < 5 mg/L measured by high-sensitivity immunoassay | 15 weeks
  Blood will be collected at baseline and during the intervention. Serum CRP concentration will be quantified using a validated high-sensitivity immunoassay (ELISA). The outcome is the proportion of participants whose CRP is < 5 mg/L during intervention. The main comparison is the between-group difference (intervention vs placebo) in the proportion meeting this threshold.
Proportion of participants with ≥50% reduction in C-reactive protein (CRP) from baseline measured by high-sensitivity immunoassay | 15 weeks
  Serum CRP will be measured at baseline and during the intervention using ELISA. The outcome is the proportion of participants who achieve ≥50% reduction in CRP compared to baseline. The primary comparison is the between-group difference (intervention vs placebo) in the percentage of participants meeting this criterion.
Proportion of participants with ≥50% reduction in stool calprotectin concentration measured by ELISA | 15 weeks
  Stool samples will be analyzed for calprotectin concentration using ELISA. The endpoint is the proportion of participants achieving a ≥50% reduction from baseline to Week 15. The between-group difference (intervention vs placebo) in the proportion of responders will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maldonado-Contreras, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMASS medical center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No